CLINICAL TRIAL: NCT02905227
Title: A Phase 1 Study of the Pulmonary Safety and Pharmacokinetics of Zolmitriptan Inhalation Powder in Chronic Smokers and People With Mild or Moderate Asthma Compared to Healthy Volunteers
Brief Title: A Study of the Pulmonary Safety and Pharmacokinetics of Zolmitriptan Inhalation Powder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIP-PK-1041
Record Dates: First submitted 2016-09-02; First posted 2016-09-19 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2017-01

CONDITIONS: Migraine
Keywords: Adult smokers; Asthma; Healthy volunteers
MeSH Terms: conditions — Migraine Disorders; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Adult Asthmatics (Experimental): Two doses of CVT-427, 2 hours apart. 3.0 mg zolmitriptan capsule administered via CVT-427 breath-actuated inhaler in adult asthmatics
  Interventions: Drug: CVT-427 (zolmitriptan inhalation powder)
- Adult Smokers (Experimental): Two doses of CVT-427, 2 hours apart. 3.0 mg zolmitriptan capsule administered via CVT-427 breath-actuated inhaler in adult smokers.
  Interventions: Drug: CVT-427 (zolmitriptan inhalation powder)
- Adult Healthy Volunteers (Experimental): Two doses of CVT-427, 2 hours apart. 3.0 mg zolmitriptan capsule administered via CVT-427 breath-actuated inhaler in adult healthy volunteers.
  Interventions: Drug: CVT-427 (zolmitriptan inhalation powder)

INTERVENTIONS:
Drug: CVT-427 (zolmitriptan inhalation powder) — Each subject received 2 self-administered doses of 3.0 mg CVT-427 (zolmitriptan inhalation powder), 2 hours apart.

SUMMARY:
This study is an open-label, parallel group study to evaluate acute pulmonary safety and Pharmacokinetics (PK) of two doses, separated by 2 hours, of CVT-427 zolmitriptan inhalation powder in three groups of adults: those with asthma, those who smoke and healthy volunteers.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate acute pulmonary safety and PK of CVT-427 zolmitriptan inhalation powder in the study populations.

ELIGIBILITY:
Inclusion Criteria:

* eligible subjects will be men or women aged 18 to 65 years inclusive;
* body mass index (BMI) 18 to 30 kg/m2;
* healthy adults must be in general good health with no clinically significant abnormalities that would affect ability to complete study.
* subjects with asthma must be non-smokers who have a forced expiratory volume in one second (FEV1) ≥ 60% of predicted for race, age, sex, and height;
* subjects who smoke must have at least a 12-month, 0.5 pack of cigarettes per day history or the equivalent consumption of cigars and a positive result for plasma cotinine.

Exclusion Criteria:

* subjects with asthma will be excluded for more than 2 hospitalizations or emergency room visits, or more than 3 courses of systemic steroids in the past 12 months or 1 course within the past 8 weeks for respiratory illness;
* asthma exacerbation within 8 weeks of before screening;
* unscheduled or urgent visit to any medical facility for asthma-related problems within 8 weeks before screening;
* history of intubation or intensive care unit admission for asthma in the past 5 years.
* Subjects who smoke will be excluded if they have intrinsic lung disease including asthma or chronic obstructive pulmonary disease (COPD) with an FEV1 of <60% of predicted and a score of ≥2 on the Medical Research Council Dsypnea Scale (MRC);
* any cardiovascular risk factor or contraindication for the use of triptans
* use of nonselective monamine oxidase inhibitors (MAOI), serotonin reuptake inhibitors (SSRIs), propranolol, or cimetidine within 4 weeks prior to the Screening Visit, or planned use during the study;
* positive serology test (hepatitis B virus surface antigen [HBsAg], hepatitis C virus [HCV] antibody, human immunodeficiency virus [HIV] 1 & 2 antibodies).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in measure of pulmonary function via Spirometry | within 1 hour prior to dose and up to 24 hours post-dose.
Maximum observed plasma drug concentration (Cmax) | up to 24 hours post-dose.
Maximum observed plasma drug concentration (tmax) | up to 24 hours post-dose.
Area under the concentration time curve over the dosing interval (AUC0-last) | up to 24 hours post-dose.

SECONDARY OUTCOMES:
Number of subjects with Adverse Events (AEs) including Serious AEs | up to 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Charles Oh, MD, Study Director — Acorda Therapeutics
Locations (3):
- United States (3):
  - Site #103, North Dartmouth, Massachusetts
  - Site #102, Lincoln, Nebraska
  - Site #101, Dallas, Texas